CLINICAL TRIAL: NCT03996603
Title: IMPLORE Study: Investigation of Microbiomes of Postmenopausal Women Looking for Outcomes and Response to Estrogen Therapy
Brief Title: Investigation of Microbiomes of Postmenopausal Women Looking for Outcomes and Response to Estrogen Therapy
Acronym: IMPLORE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Kyle P Norris, MD, Instructor Fellow, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-300002968
Record Dates: First submitted 2019-06-11; First posted 2019-06-25 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Female Urogenital Diseases; Vaginal Atrophy; Postmenopausal Atrophic Vaginitis; Genitourinary Disease; Postmenopausal Symptoms
Keywords: Genitourinary Syndrome of Menopause; Vaginal Atrophy; Vaginal Estrogen Therapy; Inflammatory Response; Microbial Colonization; Urinary Microbiome; Vaginal Microbiome; Rectal Microbiome; Conjugated Estrogen Cream
MeSH Terms: conditions — Female Urogenital Diseases; Atrophic Vaginitis; Urogenital Diseases; Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Conjugated Estrogens Cream (Experimental): 0.625mg/1g cream, 1g applied vaginally nightly for 2 weeks then 2x/week for 8 weeks
  Interventions: Drug: Conjugated Estrogens Cream
- Control Cohort (No Intervention): No intervention will be given.

INTERVENTIONS:
Drug: Conjugated Estrogens Cream — 0.625mg/1g cream, 1g applied vaginally nightly for 2 weeks then 2x/week for 8 weeks
  Other Names: Premarin Vaginal Cream
  Arms: Conjugated Estrogens Cream

SUMMARY:
In this proposed pilot study, 16S ribosomal RNA (rRNA) gene sequencing will be used in the analysis of bacterial communities (microbiomes) in postmenopausal women with vulvovaginal atrophy (VVA) before and after eight weeks of vaginal estrogen use. The investigators plan to characterize the composition and dynamics of the microbiomes of the vagina, bladder, and rectum for quantitative and qualitative changes in the distribution of operational taxonomic units (OTUs) before and after eight weeks of local vaginal estrogen therapy. Although the vagina, bladder, and gut microbiomes have been increasingly independently studied, less is known about the interactions of the bacterial communities among the three environments as well as the dynamic relationship with menopausal status and vaginal estrogen therapy and the investigators seek to elucidate these relationships further.

DETAILED DESCRIPTION:
This is an open-label pilot study of vaginal estrogen therapy in postmenopausal participants with vulvovaginal atrophy. The investigators seek to evaluate the effects of vaginal estrogen therapy on the vaginal, urinary, and rectal bacterial communities (microbiomes) and assess the (i) quantitative change in relative abundance of Lactobacillus among the community composition of bacteria in the vagina, and (ii) to evaluate the vaginal maturation index (VMI), vaginal pH, and vaginal inflammatory biomarkers: IL-1B, IL-4, IL-6, IL-8, IL-10, TNF-a, MCP-1, GM-CSF (IL - Interleukin, TNF - tumor necrosis factor, MCP - monocyte chemoattractant protein, GM - granulocyte macrophage, CSF - colony stimulating factor) and correlate any notable changes with changes noted in the vaginal microbiome, and (iii and iv) observe for quantitative and qualitative changes in the distribution of operational taxonomic units (OTUs) among the bladder and rectal microbiomes. These changes will also be compared to the results yielded from the vaginal microbiome analysis. Additionally the investigators will assess for quantitative changes in the bladder and rectal inflammatory biomarkers (IL-1B, IL-4, IL-6, IL-8, IL-10, TNF-a, MCP-1, GM-CSF) and correlate these findings with any notable changes in the bladder and rectal microbiomes. Furthermore, changes in these biomarkers will be compared with the data (inflammatory and microbial) yielded from vaginal sampling. Bio-specimens and patient questionnaires will be assessed at baseline and again after eight weeks of vaginal estrogen therapy.

20 participants will receive the intervention (vaginal estrogen therapy) for 8 weeks. 5 participants who meet the same inclusion/exclusion criteria will not receive the intervention and will be sampled at the same time points. The additional 5 participants are intended to serve as a control cohort to demonstrate stability of the microbiome over the study period. The 5 participants may be compared to the 20 participants receiving therapy but that is not part of the primary or secondary outcomes.

The investigators believe that examining the dynamic relationships of the genitourinary-rectal region is innovative and vital to validating the investigator's understanding and assumptions of the pathophysiology and treatment approaches of this disorder.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal with vulvovaginal atrophy
* Age ≥55 years old and a screening vaginal pH of ≥5.
* Without menses for ≥12 months.
* No uterovaginal or vaginal vault prolapse beyond the hymen.
* No estrogen replacement within the last month (may come off current treatment, i.e. wash out, to join the study)

Exclusion Criteria:

* Patients with BMI >35kg/m2
* Any patients with infections requiring antibiotic or antifungal therapy during the study period.
* Study patients may not use any vaginal suppositories, douches, or vaginal hygiene wipes within the month preceding enrollment. For patients already on hormone therapy, will be allowed to undergo a "wash out" period of estrogen or progesterone products for one month prior to enrollment.
* Additional exclusions included patients with systemic conditions requiring immunosuppressive drugs, currently receiving chemotherapy, or history of pelvic radiation.
* Any patients with contraindications to vaginal estrogen therapy including: vaginal bleeding of unknown etiology; known, suspected, or history of breast cancer or estrogen-dependent neoplasia; active DVT, PE, or h/o these conditions; active arterial thromboembolic disease (ie. stroke or MI) or h/o of these; known liver disease or thrombophilic disorders.
* Current tobacco use.
* Allergy to Premarin® or its constituents.
* Concurrent use of steroid creams for other indications (ie. lichen sclerosis)

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle P Norris, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conjugated Estrogens Cream | Control Cohort
Started | 20 | 5
Completed | 16 | 5
Not Completed | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conjugated Estrogens Cream | Control Cohort | Total
Number analyzed (Participants) | 20 | 5 | 25
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 65.5 [57 to 71] | 71 [61 to 77] | 66 [57 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 5 | 25
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 14 | 3 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 5 | 25
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 27.3 [23.8 to 30.9] | 30.9 [21 to 31.5] | 27.3 [22.4 to 31.7]
Parity [Median (Inter-Quartile Range); unit: births] | 2 [1.5 to 2] | 2 [1 to 2] | 2 [1 to 2]
Spontaneous Vaginal Delivery [Median (Inter-Quartile Range); unit: deliveries] | 2 [0.5 to 2] | 1 [1 to 2] | 2 [0.5 to 2]
Hysterectomy [Count of Participants; unit: Participants] | 10 | 2 | 12
Prior Prolapse Surgery [Count of Participants; unit: Participants] | 2 | 2 | 4
Prior SUI Surgery [Count of Participants; unit: Participants] | 2 | 1 | 3
Recurrent UTIs [Count of Participants; unit: Participants] | 2 | 0 | 2
Diabetes Mellitus [Count of Participants; unit: Participants] | 4 | 0 | 4
Currently on OAB/UUI Medication(s) [Count of Participants; unit: Participants] | 3 | 2 | 5
Currently Sexually Active [Count of Participants; unit: Participants] | 12 | 2 | 14
Vaginal pH [Median (Inter-Quartile Range); unit: pH] | 6.8 [6.5 to 7.5] | 7 [5.5 to 8] | 7 [6.25 to 7.5]
Vaginal Maturation Index [Median (Inter-Quartile Range); unit: units on a scale] — The maturation value (MV) is calculated with the following formula: MV = % surface cells + (0.5 × % intermediate cells)
  units on a scale | 37.5 [10 to 50] | 40 [35 to 50] | 40 [10 to 50]

OUTCOME MEASURES:

1. Primary Outcome: Quantitative Change in Relative Abundance of Lactobacillus Among the Community Composition of Bacteria in the Vagina
Description: The relative abundance of the Lactobacillus genus, as measured by 16S ribosomal RNA (rRNA) gene sequencing, is the proportion of Lactobacillus genus among the total vaginal microbiome. After analysis of the gene sequencing, the total yield of bacteria at the genus level equals 1.
  The quantitative change in relative abundance of Lactobacillus among the community composition of bacteria in the vagina will be assessed from baseline to 8 weeks. The investigators hypothesize that a pre-specified statistically significant quantitative increase in the relative abundance of Lactobacillus will be seen among the participants that receive treatment.
Time Frame: Baseline, 8 weeks
Measure: Median (Inter-Quartile Range); unit: Relative abundance
Arm/Group | Conjugated Estrogens Cream | Control Cohort
Number analyzed (Participants) | 20 | 5
Relative abundance
  Baseline | 0.07 [0.02 to 0.14] | 0.09 [0.03 to 0.45]
  8 weeks | 0.12 [0.06 to 0.96] | 0.04 [0.04 to 0.2]

2. Secondary Outcome: Change in Vaginal Maturation Index (VMI)
Description: The maturation value (MV) is calculated with the following formula: MV = % surface cells + (0.5 × % intermediate cells).
  The outcome data is reported as the delta change from baseline to 8 weeks.
  The data for the primary outcome has been entered using the "measure type - NUMBER" because the outcome is a delta or change in the vaginal maturation index.
Time Frame: Baseline, 8 weeks
Measure: Median (Inter-Quartile Range); unit: Change in vaginal maturation index value
Arm/Group | Conjugated Estrogens Cream | Control Cohort
Number analyzed (Participants) | 20 | 5
Change in vaginal maturation index value
  Baseline | 35 [10 to 47.5] | 42.5 [17.5 to 50]
  8 weeks | 60 [50 to 65] | 47.5 [45 to 52.5]

3. Secondary Outcome: Change in Vaginal pH
Description: Change in the vaginal pH from baseline to 8 weeks
Time Frame: Baseline, 8 weeks
Measure: Median (Inter-Quartile Range); unit: Vaginal pH
Arm/Group | Conjugated Estrogens Cream | Control Cohort
Number analyzed (Participants) | 20 | 5
Vaginal pH
  Baseline | 7.25 [6.5 to 7.5] | 7 [5.5 to 8.0]
  8 weeks | 5 [4.5 to 5.5] | 7 [5.5 to 7.5]

4. Secondary Outcome: Vaginal Inflammatory Biomarkers: IL-1B, IL-4, IL-6, IL-8, IL-10, TNF-a, MCP-1, GM-CSF
Description: Change in the vaginal inflammatory biomarkers: IL-1B, IL-4, IL-6, IL-8, IL-10, TNF-a, MCP-1, GM-CSF from baseline to 8 weeks
Time Frame: Baseline, 8 weeks
Population: Only one specimen resulted in a value for IL-10 post-treatment.
Measure: Median (Inter-Quartile Range); unit: pg/mg
Arm/Group | Conjugated Estrogens Cream | Control Cohort
Number analyzed (Participants) | 20 | 5
pg/mg
  IL-1b BASELINE | 44.4 [5.9 to 84.9] | 132.9 [28.8 to 236.9]
  IL-1b 8 WEEKS | 10.8 [4.0 to 26.0] | 373.6 [10.2 to 737.1]
  IL-4 BASELINE | 10.0 [5.3 to 23.1] | 18.1 [2.3 to 33.8]
  IL-4 8 WEEKS | 2.1 [1.3 to 4.2] | 11.1 [5.0 to 17.2]
  IL-8 BASELINE | 3158.2 [1956.2 to 8087.5] | 3724.3 [2254.4 to 5194.2]
  IL-8 8 WEEKS | 757.5 [260.0 to 1980.3] | 7941.0 [2247.8 to 13643.2]
  IL-10 BASELINE | 22.5 [14.9 to 38.2] | 12.7 [1.7 to 22.1]
  IL-10 8 WEEKS: number analyzed (Participants) | 1 | 5
  IL-10 8 WEEKS | 640.7 [NA to NA] — Only one specimen resulted a value for IL-10 post treatment. | 7.0 [5.1 to 14.3]
  TNF-a BASELINE | 9.3 [8.9 to 56.9] | 11.6 [6.1 to 39.7]
  TNF-a 8 WEEKS | 7.1 [6.5 to 10.1] | 12.0 [7.2 to 30.5]
  MCP-1 BASELINE | 102.5 [22.1 to 232.1] | 29.1 [24.4 to 186.7]
  MCP-1 8 WEEKS | 6.7 [3.3 to 31.3] | 59.0 [19.8 to 79.1]

5. Other Pre Specified Outcome: Quantitative and Qualitative Changes in the Distribution of Operational Taxonomic Units (OTUs) in the Bladder Microbiome.
Description: Quantitative and qualitative changes in the distribution of operational taxonomic units (OTUs) from baseline to 8 weeks.
Time Frame: Baseline, 8 weeks
Population: There was only one participant and there was no range.
Arm/Group | Conjugated Estrogens Cream | Control Cohort
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Quantitative and Qualitative Changes in the Distribution of Operational Taxonomic Units (OTUs) in the Rectal Microbiome.
Description: Quantitative and qualitative changes in the distribution of operational taxonomic units (OTUs) from baseline to 8 weeks.
Time Frame: Baseline, 8 weeks
Population: This data was never collected.
Arm/Group | Conjugated Estrogens Cream | Control Cohort
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Bladder Inflammatory Biomarkers (IL-1B, IL-4, IL-6, IL-8, IL-10, TNF-a, MCP-1, GM-CSF)
Description: Change in the concentration of bladder inflammatory biomarkers: IL-1B, IL-4, IL-6, IL-8, IL-10, TNF-a, MCP-1, GM-CSF from baseline to 8 weeks
Time Frame: Baseline, 8 weeks
Population: This data was never collected.
Arm/Group | Conjugated Estrogens Cream | Control Cohort
Number analyzed (Participants) | 0 | 0

8. Other Pre Specified Outcome: Rectal Inflammatory Biomarkers (IL-1B, IL-4, IL-6, IL-8, IL-10, TNF-a, MCP-1, GM-CSF)
Description: Change in the concentration of rectal inflammatory biomarkers: IL-1B, IL-4, IL-6, IL-8, IL-10, TNF-a, MCP-1, GM-CSF from baseline to 8 weeks
Time Frame: Baseline, 8 weeks
Population: This data was never collected.
Arm/Group | Conjugated Estrogens Cream | Control Cohort
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Conjugated Estrogens Cream | Control Cohort
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/5
Other Adverse Events (participants affected / at risk) | 0/20 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT03996603/Prot_SAP_000.pdf